CLINICAL TRIAL: NCT02711033
Title: Laparoscopic-assisted Total Gastrectomy Versus Open Total Gastrectomy With Spleen-preserving Splenic Hilum Lymph Nodes Dissection for Advanced Proximal Gastric Cancer: A Randomized Controlled Trial
Brief Title: Laparoscopic-assisted Total Gastrectomy Versus Open Total Gastrectomy With Splenic Hilum Lymph Nodes Dissection
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Guangdong Provincial Hospital of Traditional Chinese Medicine (Other)
Responsible Party: Principal Investigator, Wei Wang, M.D., PhD., Guangdong Provincial Hospital of Traditional Chinese Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GDPHCM-GI-01
Record Dates: First submitted 2016-03-09; First posted 2016-03-17 (Estimated); Last update posted 2017-04-10 (Actual); Status verified 2017-04

CONDITIONS: Gastric Cancer; Splenic Hilum Lymph Nodes Dissection; Total Gastrectomy
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Laparoscopic-assisted total gastrectomy (Experimental): Patients including in the laparoscopic-assisted total gastrectomy (LATG) group will undergo LATG with spleen-preserving splenic hilum lymph nodes dissection.
  Interventions: Procedure: Laparoscopic-assisted total gastrectomy
- Open total gastrectomy (Active Comparator): Patients who are included in the open total gastrectomy (OTG) group will OTG with spleen-preserving splenic hilum lymph nodes dissection.
  Interventions: Procedure: Open total gastrectomy

INTERVENTIONS:
Procedure: Laparoscopic-assisted total gastrectomy — When patients with advanced proximal gastric cancer are randomized in the laparoscopic-assisted total gastrectomy (LATG) group, they will received LATG with spleen-preserving splenic hilum lymph nodes dissection.
  Other Names: LATG
  Arms: Laparoscopic-assisted total gastrectomy
Procedure: Open total gastrectomy — When patients with advanced proximal gastric cancer are randomized in the open total gastrectomy (OTG) group, they will received OTG with spleen-preserving splenic hilum lymph nodes dissection.
  Other Names: OTG
  Arms: Open total gastrectomy

SUMMARY:
This study investigates the safety and feasibility of laparoscopic-assisted total gastrectomy with spleen-preserving splenic hilum lymph node dissection for proximal advanced gastric cancer and compares the early results of this procedure with open total gastrectomy.

DETAILED DESCRIPTION:
For advanced proximal gastric cancer, total gastrectomy with D2 lymphadenectomy is the standard surgical therapy. Apparently, lymph nodes (LNs) dissection along the splenic artery (No.11) and the splenic hilum (No.10) is recommended by the Japanese Gastric Cancer Treatment Guidelines. Nevertheless, complete removal of the No. 10 and No. 11d LNs is technically challenging due to the tortuous splenic vessels and the high possibility of injury to the parenchyma of the spleen and pancreas. Recently, the application of minimally invasive surgery for advanced gastric cancer is gaining popularity. However, laparoscopic-assisted total gastrectomy (LATG) with standard D2 lymphadenectomy was still not widely performed, because pancreas- and spleen-preserving splenic hilum lymph node dissection were mainly challenging manipulations for laparoscopic surgeons. Herein, we aim to investigate the safety and feasibility of LATG with spleen-preserving splenic hilum lymph node dissection for proximal advanced gastric cancer and compares the early results of this procedure with open total gastrectomy (OTG).

ELIGIBILITY:
Inclusion Criteria:

* Patient with advanced proximal gastric cancer （T2-T4a,N0-N3,M0）
* Informed consent
* Eastern Cooperative Oncology Group (ECOG): 0 ot 1
* American Society of Anesthesiologists （ASA） score: Ⅰto Ⅲ

Exclusion Criteria:

* Pregnancy or female in suckling period
* Contraindication to general anesthesia (severe cardiac and/or pulmonary disease)
* Severe mental disease
* Emergency operation due to complication (bleeding, perforation or obstruction) caused by primary tumor
* Body mass index (BMI) > 30 kg/m2

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Estimated)
Dates: Start 2015-10; Primary Completion 2018-10 (Estimated); Study Completion 2019-04 (Estimated)

PRIMARY OUTCOMES:
Early complication rate | 30 days
  The early complication rate is defined as the event observed during operation and within 30 days after surgery.

SECONDARY OUTCOMES:
Operative time | Intraoperative
Time of splenic hilum lymph nodes dissection | Intraoperative
Operative blood loss | Intraoperative
  It will be assessed with the unit of "ml".
Incision length | 7 days
Number of total lymph nodes harvested | 7 days
Number of group No.10 lymph nodes harvested | 7 days
Number of lymph nodes posterior to splenic vessel | 7 days
Poster-operative recovery course | 30 days
  Time to first ambulation, flatus, liquid diet and duration of hospital stay are used to assess the postoperative recovery course.
3-year disease free survival rate | 3 years
5-year overall survival rate | 5 years
Metastasis rate of lymph nodes posterior to splenic vessel | 7 days

CONTACTS AND LOCATIONS:
Overall Officials: Wei Wang, M.D., PH.D., Principal Investigator — Guangdong Province Hospital of Chinese Medicine, the Second Affiliated Hospital of Guangzhou University of Chinese Medicine
Locations (1):
- Guangdong Province Hospital of Chinese Medicine, the Second Affiliated Hospital of Guangzhou University of Chinese Medicine, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No